CLINICAL TRIAL: NCT03188692
Title: Phase 3 Study of BK1310 Intramuscular Injection in Healthy Infants
Brief Title: Safety and Efficacy of BK1310 Intramuscular Injection in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Collaborators: The Research Foundation for Microbial Diseases of Osaka University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BK1310-J02
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Immunization
Keywords: Haemophilus influenza type b; Adsorbed Diphtheria-Purified Pertussis-Tetanus-Inactivate; poliovirus combined vaccine; Hib; DPT-IPV; Intramuscular
MeSH Terms: conditions — Haemophilus Infections | interventions — Vaccines, Combined

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BK1310 (Experimental)
  Interventions: Biological: DPT-IPV-Hib (Combined Vaccine)

INTERVENTIONS:
Biological: DPT-IPV-Hib (Combined Vaccine) — 0.5mL, intramuscular injection, 3 times with the 3-8weeks intervals then an additional injection after 6-13 months.
  Other Names: BK1310

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of an intramuscular injection of BK1310 in healthy infants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants aged ≥2 and <43 months at the first vaccination of the study drug (recommended: ≥2 and <7 months). Those who are applicable of the following conditions must be carefully observed before the enrollment: infants with known underlying disease such as cardiovascular disease, renal disease, hepatic disease, blood dyscrasia, respiratory disease or developmental disorder. Infants who developed fever within 2 days after any previous vaccination. Infants with history of convulsions.
* Written informed consent is obtained from a legal guardian (parent)

Exclusion Criteria:

* With past diagnosis of immunodeficiency or currently under immunosuppressive treatment
* Have close relatives (the third degree of kinship) diagnosed with congenital immunodeficiency
* Possibility of anaphylaxis due to food or pharmaceuticals
* With diagnosis of thrombocytopenia and/or coagulopathy or currently under treatment of the antiplatelet agents and/or anticoagulant agents.
* With experience of Hib infection, diphtheria, pertussis, tetanus or acute poliomyelitis
* With experience of Hib, diphteria, pertussis, tetanus or polio vaccination.
* Administered a live vaccine within 27 days before the first vaccination of the study drug, or inactivated vaccine or toxoid within 6 days before vaccination
* Administered transfusion, immunosuppressant (excluding drugs for external use), or immunoglobulin formulation
* Administered corticosteroid 2 mg/kg per day or more as prednisolone (excluding drugs for external use)
* Participated in other studies within 12 weeks before obtaining consent
* With the gestational age <37 weeks or weighed less than 2500 grams at birth.
* Considered to be not eligible by the principal investigators (sub-investigators) of the enrollment.

Ages: 2 Months to 43 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2018-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (3):
- Japan (3):
  - Investigational site 1, Chiba
  - Investigational site 2, Tokyo
  - Investigational site 3, Tokyo

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BK1310
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | BK1310
Number analyzed (Participants) | 33
Age, Customized [Count of Participants; unit: Participants]
  >=2 and <3 months | 27
  >=3 months | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian (Japanese) | 33

OUTCOME MEASURES:

1. Primary Outcome: Antibody Prevalence Rate Against Anti-PRP With 1 μg/mL or Higher, Diphtheria Toxin, Pertussis, Tetanus Toxin, and Polio Virus, Defined as the Percentage of Participants With the Antibody Against Anti-PRP
Description: Antibody prevalence rate is defined as the percentage of participants whose criteria of each antibody titer: Anti-diphtheria antibody concentrations: >=0.1 IU/mL, Anti-PT antibody concentrations: >=10.0 EU/mL, Anti-FHA antibody concentrations: >=10.0 EU/mL, Anti-tetanus antibody concentrations: >=0.01 IU/mL, Anti-poliovirus serotype 1,2 and 3 antibody titers (fold) >=8
Time Frame: 4 weeks after the primary immunization (Visit 4)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BK1310
Number analyzed (Participants) | 33
percentage of participants
  Antibody prevalence rate against anti-PRP with 1 μg/mL or higher | 97.0 [84.2 to 99.9]
  Antibody prevalence rate against diphtheria toxin | 93.9 [79.8 to 99.3]
  Antibody prevalence rate against pertussis （PT） | 100.0 [89.4 to 100.0]
  Antibody prevalence rate against pertussis (FHA) | 97.0 [84.2 to 99.9]
  Antibody prevalence rate against tetanus toxin | 100.0 [89.4 to 100.0]
  Antibody prevalence rate against polio virus serotype 1 | 100.0 [89.4 to 100.0]
  Antibody prevalence rate against polio virus serotype 2 | 100.0 [89.4 to 100.0]
  Antibody prevalence rate against polio virus serotype 3 | 100.0 [89.4 to 100.0]

2. Secondary Outcome: Anti-PRP Antibody Prevalence Rate With 0.15 μg/mL or Higher, Defined as the Percentage of Participants With the Anti-PRP Antibody
Time Frame: 4 weeks after the primary immunization (Visit 4)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BK1310
Number analyzed (Participants) | 33
percentage of participants | 100.0 [89.4 to 100.0]

3. Secondary Outcome: Geometric Mean Antibody Titer of Anti-PRP Antibody
Time Frame: 4 weeks after the primary immunization (Visit 4)
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | BK1310
Number analyzed (Participants) | 33
µg/mL | 13.522 [8.628 to 21.192]

4. Secondary Outcome: Anti-PRP Antibody Prevalence Rate With 1 μg/mL or Higher, Defined as the Percentage of Participants With the Anti-PRP Antibody
Time Frame: 4 weeks after the booster dose (Visit 6)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BK1310
Number analyzed (Participants) | 33
percentage of participants | 100.0 [89.4 to 100.0]

5. Secondary Outcome: Anti-PRP Antibody Prevalence Rate With 0.15 μg/mL or Higher, Defined as the Percentage of Participants With the Anti-PRP Antibody
Time Frame: 4 weeks after the booster dose (Visit 6)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BK1310
Number analyzed (Participants) | 33
percentage of participants | 100.0 [89.4 to 100.0]

6. Secondary Outcome: Geometric Mean Antibody Titer of Anti-PRP Antibody
Time Frame: 4 weeks after the booster dose (Visit 6)
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | BK1310
Number analyzed (Participants) | 33
µg/mL | 28.509 [20.866 to 38.952]

7. Secondary Outcome: Geometric Mean Antibody Titer Against Diphtheria Toxin
Time Frame: 4 weeks after the primary immunization (Visit 4)
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BK1310
Number analyzed (Participants) | 33
IU/mL | 1.0818 [0.7157 to 1.6352]

8. Secondary Outcome: Geometric Mean Antibody Titer Against Pertussis （PT）
Time Frame: 4 weeks after the primary immunization (Visit 4)
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | BK1310
Number analyzed (Participants) | 33
EU/mL | 128.03 [106.09 to 154.51]

9. Secondary Outcome: Geometric Mean Antibody Titer Against Pertussis （FHA）
Time Frame: 4 weeks after the primary immunization (Visit 4)
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | BK1310
Number analyzed (Participants) | 33
EU/mL | 53.64 [44.01 to 65.40]

10. Secondary Outcome: Geometric Mean Antibody Titer Against Tetanus Toxin
Time Frame: 4 weeks after the primary immunization (Visit 4)
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BK1310
Number analyzed (Participants) | 33
IU/mL | 0.3068 [0.2091 to 0.4502]

11. Secondary Outcome: Fold Change in Geometric Mean Antibody Titer Against Polio Virus
Time Frame: Baseline and 4 weeks after the primary immunization (Visit 4)
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | BK1310
Number analyzed (Participants) | 33
fold change
  Geometric mean antibody titer against polio virus serotype 1 | 551.06 [348.74 to 870.74]
  Geometric mean antibody titer against polio virus serotype 2 | 1510.29 [1046.26 to 2180.11]
  Geometric mean antibody titer against polio virus serotype 3 | 1290.16 [937.99 to 1774.55]

12. Secondary Outcome: Antibody Prevalence Rate Against Diphtheria Toxin, Pertussis, Tetanus Toxin, and Polio Virus, Defined as the Percentage of Participants With the Antibody Against Diphtheria Toxin, Pertussis, Tetanus Toxin, and Polio Virus
Description: as for outcome 1
Time Frame: 4 weeks after the booster dose (Visit 6)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BK1310
Number analyzed (Participants) | 33
percentage of participants
  Antibody prevalence rate against diphtheria toxin | 100.0 [89.4 to 100.0]
  Antibody prevalence rate against pertussis （PT） | 100.0 [89.4 to 100.0]
  Antibody prevalence rate against pertussis （FHA） | 100.0 [89.4 to 100.0]
  Antibody prevalence rate against tetanus toxin | 100.0 [89.4 to 100.0]
  Antibody prevalence rate against polio virus serotype 1 | 100.0 [89.4 to 100.0]
  Antibody prevalence rate against polio virus serotype 2 | 100.0 [89.4 to 100.0]
  Antibody prevalence rate against polio virus serotype 3 | 100.0 [89.4 to 100.0]

13. Secondary Outcome: Geometric Mean Antibody Titer Against Diphtheria Toxin
Time Frame: 4 weeks after the booster dose (Visit 6)
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BK1310
Number analyzed (Participants) | 33
IU/mL | 9.6485 [7.2551 to 12.8316]

14. Secondary Outcome: Geometric Mean Antibody Titer Against Pertussis （PT）
Time Frame: 4 weeks after the booster dose (Visit 6)
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | BK1310
Number analyzed (Participants) | 33
EU/mL | 173.17 [140.90 to 212.84]

15. Secondary Outcome: Geometric Mean Antibody Titer Against Pertussis （FHA）
Time Frame: 4 weeks after the booster dose (Visit 6)
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | BK1310
Number analyzed (Participants) | 33
EU/mL | 114.19 [89.14 to 146.28]

16. Secondary Outcome: Geometric Mean Antibody Titer Against Tetanus Toxin
Time Frame: 4 weeks after the booster dose (Visit 6)
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | BK1310
Number analyzed (Participants) | 33
IU/mL | 1.8293 [1.2107 to 2.7640]

17. Secondary Outcome: Fold Change in Geometric Mean Antibody Titer Against Polio Virus
Time Frame: Baseline and 4 weeks after the primary immunization (Visit 6)
Measure: Geometric Mean (95% Confidence Interval); unit: fold change
Arm/Group | BK1310
Number analyzed (Participants) | 33
fold change
  Geometric mean antibody titer against polio virus serotype 1 | 1642.66 [1162.23 to 2321.68]
  Geometric mean antibody titer against polio virus serotype 2 | 8910.01 [6877.46 to 11543.27]
  Geometric mean antibody titer against polio virus serotype 3 | 5000.58 [3839.01 to 6513.60]

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 year
Arm/Group | BK1310
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 2/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BK1310 (N=33)
Bronchiolitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Exanthema subitum (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BK1310 (N=33)
Constipation (Gastrointestinal disorders) | 2
Crying (General disorders) | 11
Injection site erythema (General disorders) | 16
Injection site induration (General disorders) | 5
Injection site swelling (General disorders) | 6
Irritability postvaccinal (General disorders) | 4
Pyrexia (General disorders) | 25
Bronchitis (Infections and infestations) | 5
Conjunctivitis (Infections and infestations) | 5
Gastroenteritis (Infections and infestations) | 5
Hand-foot-and-mouth disease (Infections and infestations) | 2
Otitis media (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 2
Viral upper respiratory tract infection (Infections and infestations) | 2
Arthropod sting (Injury, poisoning and procedural complications) | 3
Decreased appetite (Metabolism and nutrition disorders) | 5
Hypersomnia (Nervous system disorders) | 10
Insomnia (Psychiatric disorders) | 7
Asthma (Respiratory, thoracic and mediastinal disorders) | 5
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 11
Asteatosis (Skin and subcutaneous tissue disorders) | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2
Eczema infantile (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-05-24): https://cdn.clinicaltrials.gov/large-docs/92/NCT03188692/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-09): https://cdn.clinicaltrials.gov/large-docs/92/NCT03188692/SAP_001.pdf